CLINICAL TRIAL: NCT02486653
Title: Pre-operative Tamsulosin for the Prevention of Post-operative Urinary Retention: a Randomized, Double-blind, Placebo-controlled Trial
Brief Title: Prevention of Post-operative Urinary Retention
Acronym: POUR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2014-1494
Record Dates: First submitted 2015-06-25; First posted 2015-07-01 (Estimated); Results first posted 2019-04-23 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Urinary Retention; Urinary Tract Infections
Keywords: tamsulosin; randomized controlled trials as topic; double-blind method; random allocation; placebos; Adrenergic alpha-Antagonists; urinary retention; urinary tract infections; urinary catheters; catheter-related infections; postoperative complications
MeSH Terms: conditions — Urinary Retention; Urinary Tract Infections; Catheter-Related Infections; Postoperative Complications | interventions — Tamsulosin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tamsulosin (Experimental)
  Interventions: Drug: Tamsulosin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tamsulosin — Tamsulosin 0.4mg capsule orally once daily, dosed 30 minutes after dinner or before bed, starting 7 days before surgery and continuing for 0-5 days postoperatively.
  Outline of schedule:
  * Day 1-7: tamsulosin 0.4mg in the evening
  * Day 8: surgery; tamsulosin 0.4mg in the evening if the subject has not yet completed the bladder management protocol
  * Day 9-14: tamsulosin 0.4mg in the evening until the subject either 1) completes the bladder management protocol (defined by two consecutive voids with post-void residual <200mL), or 2) has an indwelling urinary catheter replaced, or 3) is discharged from the hospital, whichever occurs first. The minimum number of total doses is 7; the maximum number of total doses is 14. The 14th dose will be the final dose regardless of bladder function.
  Other Names: Flomax
  Arms: Tamsulosin
Drug: Placebo — Placebo capsule orally once daily, dosed 30 minutes after dinner or before bed, starting 7 days before surgery and continuing for 0-5 days postoperatively.
  Outline of schedule:
  * Day 1-7: placebo in the evening
  * Day 8: surgery; placebo in the evening if the subject has not yet completed the bladder management protocol
  * Day 9-14: placebo in the evening until the subject either 1) completes the bladder management protocol (defined by two consecutive voids with post-void residual <200mL), or 2) has an indwelling urinary catheter replaced, or 3) is discharged from the hospital, whichever occurs first. The minimum number of total doses is 7; the maximum number of total doses is 14. The 14th dose will be the final dose regardless of bladder function.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if tamsulosin ("FLOMAX") is effective in preventing post-operative urinary retention following abdominal surgery. Post-operative urinary retention is a common post-operative complication, occurring in up to 30% of patients undergoing abdominal surgery. It can be described as the inability to initiate urination or properly empty one's bladder following surgery. It is usually self-limited, but it requires the use of catheterization to empty the bladder in order to prevent further injury to the bladder or kidneys and to relief the discomfort of a full bladder. Tamsulosin is a medication that is commonly used in men with urinary symptoms related to an enlarged prostate. There is some evidence to suggest that it may also potentially be beneficial for preventing post-operative urinary retention. Therefore, in this research study, subjects scheduled for abdominal surgery will be randomly assigned to take either tamsulosin once-daily or placebo once-daily for one week leading up to surgery, and up to several days after surgery. Urinary function will be assessed and compared between these two treatments. The hypothesis is that tamsulosin will reduce the rate of postoperative urinary retention compared to placebo.

DETAILED DESCRIPTION:
Postoperative urinary retention (POUR) complicates up to 30% of general abdominal operations. It results in patient discomfort, embarrassment, interference with therapies, and significant nursing burden. More importantly, urinary retention necessitates use of intermittent catheterization or placement of an indwelling urinary catheter, which exposes the patient to an increased risk of urinary tract infection (UTI), urethral injury, and potentially increased hospital length of stay and cost. For these reasons, a safe and effective intervention for preventing POUR would be highly valuable. Despite such a need, no contemporary studies exist evaluating medications that can be used to prevent POUR in broad general surgery populations. To address this gap, the investigators have designed a prospective, randomized, double-blind, placebo-controlled trial to test the hypothesis that preoperative loading with tamsulosin will prevent POUR in patients undergoing elective, inpatient complex intra-abdominal surgery and thereby lead to improved short-term outcomes.

Tamsulosin is a safe and widely-used selective alpha-1-A adrenergic blocker commonly used for the treatment of lower urinary tract symptoms in men with benign prostatic hypertrophy. It has also been shown to have some benefit in reducing POUR and need for catheterization in men undergoing inguinal hernia repair and other outpatient urologic procedures. This study is a randomized, double-blind, placebo-controlled trial in which patients scheduled for inpatient complex intra-abdominal surgery will be randomized to receive either tamsulosin or placebo for 7 days pre-operatively, and up to several days post-operatively, and then rates of POUR will be compared between the two groups (Aim 1). A retrospective analysis of the data will be used to identify risk factors for POUR and subgroups of patients that would derive the greatest benefit from preoperative tamsulosin (Aim 2). Furthermore, short-term outcomes, including rate of urinary tract infection (UTI) and hospital length of stay, will be compared between the tamsulosin and placebo groups (Aim 3).

Enrolled subjects will be randomized using a blocked, stratified randomization process to either tamsulosin or placebo. Stratification variables include gender, pelvic vs non-pelvic surgery, and International Prostate Symptom Score (IPSS) survey results (which is a measure of baseline lower urinary tract symptoms). After a 7-day treatment period, subjects will undergo surgery as scheduled, and then the assigned treatment will be continued for up to a total of 14 days until the subject either has return of normal voiding function, has required replacement of an indwelling urinary catheter, or is discharged from the hospital.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking
* Able to provide informed consent
* Scheduled to undergo an elective, complex intra-abdominal operation with a planned postoperative inpatient stay of at least 1 night

Exclusion Criteria:

* Less than age 18
* Allergy or contraindication to tamsulosin
* Serious sulfa allergy
* Current use of alpha blocker (alfuzosin, doxazosin, prazosin, silodosin, terazosin, verapamil, tamsulosin) or oral alpha agonist (midodrine), or initiation of one of these medications during the intervention phase of the study will result in subject withdrawal from the study
* Current warfarin use
* Pre-existing indwelling urinary catheter, suprapubic catheter, or urostomy
* End stage renal disease or dialysis-dependence
* Sitting systolic blood pressure in the upper extremity of less than 100mm Hg at time of eligibility screening
* Presence of orthostatic hypotension at the time of eligibility screening (orthostatic hypotension is defined as a drop in systolic blood pressure of 20mm Hg from sitting to standing, or drop in diastolic BP of 10 mm Hg from sitting to standing after 2-3 minutes of standing after being in a sitting position)
* Anticipated inability to take oral medications on post-operative day #0
* Anticipated requirement for indwelling urinary catheter beyond post-operative day #2
* Non-English speaking
* Pregnant or breast-feeding
* Unwillingness to answer all 7 questions on the IPSS (International Prostate Symptom Score) survey
* Lacking capacity to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2018-04-01 (Actual); Study Completion 2018-05-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Evie H Carchman, MD, Principal Investigator — University of Wisconsin - Madison School of Medicine and Public Health
Locations (1):
- University of Wisconsin Hospital and Clinics, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Buckley BS, Lapitan MC. Drugs for treatment of urinary retention after surgery in adults. Cochrane Database Syst Rev. 2010 Oct 6;2010(10):CD008023. doi: 10.1002/14651858.CD008023.pub2. PMID 20927768
- [Background] Choi S, Awad I. Maintaining micturition in the perioperative period: strategies to avoid urinary retention. Curr Opin Anaesthesiol. 2013 Jun;26(3):361-7. doi: 10.1097/ACO.0b013e32835fc8ba. PMID 23492981
- [Background] Lo E, Nicolle LE, Coffin SE, Gould C, Maragakis LL, Meddings J, Pegues DA, Pettis AM, Saint S, Yokoe DS. Strategies to prevent catheter-associated urinary tract infections in acute care hospitals: 2014 update. Infect Control Hosp Epidemiol. 2014 May;35(5):464-79. doi: 10.1086/675718. No abstract available. PMID 24709715
- [Background] Hollingsworth JM, Rogers MA, Krein SL, Hickner A, Kuhn L, Cheng A, Chang R, Saint S. Determining the noninfectious complications of indwelling urethral catheters: a systematic review and meta-analysis. Ann Intern Med. 2013 Sep 17;159(6):401-10. doi: 10.7326/0003-4819-159-6-201309170-00006. PMID 24042368
- [Background] O'Leary MP. Tamsulosin: current clinical experience. Urology. 2001 Dec;58(6 Suppl 1):42-8; discussion 48. doi: 10.1016/s0090-4295(01)01346-2. PMID 11750250
- [Background] Madani AH, Aval HB, Mokhtari G, Nasseh H, Esmaeili S, Shakiba M, Shakiba RS, Seyed Damavand SM. Effectiveness of tamsulosin in prevention of post-operative urinary retention: a randomized double-blind placebo-controlled study. Int Braz J Urol. 2014 Jan-Feb;40(1):30-6. doi: 10.1590/S1677-5538.IBJU.2014.01.05. PMID 24642148
- [Background] Narayan P, Tewari A. A second phase III multicenter placebo controlled study of 2 dosages of modified release tamsulosin in patients with symptoms of benign prostatic hyperplasia. United States 93-01 Study Group. J Urol. 1998 Nov;160(5):1701-6. PMID 9783935
- [Background] Lepor H. Phase III multicenter placebo-controlled study of tamsulosin in benign prostatic hyperplasia. Tamsulosin Investigator Group. Urology. 1998 Jun;51(6):892-900. doi: 10.1016/s0090-4295(98)00126-5. PMID 9609623
- [Background] Pummangura N, Kochakarn W. Efficacy of tamsulosin in the treatment of lower urinary tract symptoms (LUTS) in women. Asian J Surg. 2007 Apr;30(2):131-7. doi: 10.1016/S1015-9584(09)60146-9. PMID 17475584
- [Background] Yaycioglu O, Altan-Yaycioglu R. Intraoperative floppy iris syndrome: facts for the urologist. Urology. 2010 Aug;76(2):272-6. doi: 10.1016/j.urology.2010.01.025. Epub 2010 Mar 28. PMID 20350754
- [Background] Chang DF, Osher RH, Wang L, Koch DD. Prospective multicenter evaluation of cataract surgery in patients taking tamsulosin (Flomax). Ophthalmology. 2007 May;114(5):957-64. doi: 10.1016/j.ophtha.2007.01.011. PMID 17467530

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began in August 2015 and continued until Feb 2018. Subjects were recruited from surgery clinics at a single university hospital.
Pre-assignment Details: Subjects were randomized within 1 month of their surgery date but >7 days prior to surgery. 7 participants were not randomized for the following reasons: 4 subjects self-withdraw prior to randomization; 3 subjects had surgery date moved up to within the 7-day window before surgery
Period: Overall Study
Arm/Group | Tamsulosin | Placebo
Started | 76 | 75
Completed | 70 | 71
Not Completed | 6 | 4
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Protocol Violation | 1 | 0
Not completed — surgery cancelled | 4 | 1

BASELINE CHARACTERISTICS:
Population: 76 subjects randomized to Tamsulosin; 4 surgery cancelled, 1 withdrew prior to starting study drug, 1 had intraoperative urethral injury precluding ability to collect outcome data, therefore analysis population was 70 subjects. 75 randomized to Placebo; 3 withdrew prior to starting study drug, 1 surgery cancelled, therefore analysis pop. was 71
Groups:
- Total: Total of all reporting groups
Arm/Group | Tamsulosin | Placebo | Total
Number analyzed (Participants) | 76 | 75 | 151
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 1
  Between 18 and 65 years | 59 | 54 | 113
  >=65 years | 16 | 21 | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.7 (15.8) | 54.5 (14.4) | 53.6 (15.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 34 | 68
  Male | 42 | 41 | 83
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 73 | 73 | 146
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 76 | 75 | 151
IPSS [Count of Participants; unit: Participants] — IPSS is the International Prostate Symptom Score. This is a validated 7-question survey that characterizes severity of lower urinary tract symptoms. The score ranges from 0-35, with high scores indicating more significant symptoms (i.e. weak stream, urinary frequency, needing to strain to begin urination, etc). This is a self-completed survey filled out by the subject. Population: These are the baseline characteristics for the subjects who completed the study (and for whom there is outcomes data). Of the 151 subjects randomized, 4 withdrew prior to starting study med, 5 had surgery cancelled, and 1 had an intraop complication precluding any collection of outcomes data, yielding a total of 141 subjects.
  Participants
    number analyzed (Participants) | 70 | 71 | 141
    Low IPSS (Score <=7) | 44 | 45 | 89
    High IPSS (Score >7) | 26 | 26 | 52
Pelvic Surgery [Count of Participants; unit: Participants] — "Pelvic Surgery" was defined as surgical procedure involving dissection/resection/anastomosis involving the rectum or pelvis. Population: These are the baseline characteristics for the subjects who completed the study (and for whom there is outcomes data). Of the 151 subjects randomized, 4 withdrew prior to starting study med, 5 had surgery cancelled, and 1 had an intraop complication precluding any collection of outcomes data, yielding a total of 141 subjects.
  Participants
    number analyzed (Participants) | 70 | 71 | 141
    Non-pelvic Surgery | 30 | 32 | 62
    Pelvic Surgery | 40 | 39 | 79
Epidural [Count of Participants; unit: Participants] — This baseline characteristic describes whether or not an epidural was used for postoperative analgesia Population: These are the baseline characteristics for the subjects who completed the study (and for whom there is outcomes data). Of the 151 subjects randomized, 4 withdrew prior to starting study med, 5 had surgery cancelled, and 1 had an intraop complication precluding any collection of outcomes data, yielding a total of 141 subjects.
  Participants
    number analyzed (Participants) | 70 | 71 | 141
    Epidural used | 25 | 16 | 41
    No epidural | 45 | 55 | 100
ASA Class [Count of Participants; unit: Participants] — American Society of Anesthesiologists (ASA) Classification characterizes baseline comorbidities of patients undergoing surgery:
  Class 1- normal healthy patient Class 2- Mild systemic disease Class 3- Severe systemic disease Population: These are the baseline characteristics for the subjects who completed the study (and for whom there is outcomes data). Of the 151 subjects randomized, 4 withdrew prior to starting study med, 5 had surgery cancelled, and 1 had an intraop complication precluding any collection of outcomes data, yielding a total of 141 subjects.
  Participants
    number analyzed (Participants) | 70 | 71 | 141
    ASA Class 1 | 3 | 1 | 4
    ASA Class 2 | 48 | 55 | 103
    ASA Class 3 | 19 | 15 | 34
Body Mass Index [Count of Participants; unit: Participants] — Population: These are the baseline characteristics for the subjects who completed the study (and for whom there is outcomes data). Of the 151 subjects randomized, 4 withdrew prior to starting study med, 5 had surgery cancelled, and 1 had an intraop complication precluding any collection of outcomes data, yielding a total of 141 subjects.
  Participants
    number analyzed (Participants) | 70 | 71 | 141
    less than 30, non-obese | 38 | 42 | 80
    greater than or equal to 30, obese | 32 | 29 | 61
History of Prior Urinary Retention [Count of Participants; unit: Participants] — Population: These are the baseline characteristics for the subjects who completed the study (and for whom there is outcomes data). Of the 151 subjects randomized, 4 withdrew prior to starting study med, 5 had surgery cancelled, and 1 had an intraop complication precluding any collection of outcomes data, yielding a total of 141 subjects.
  Participants
    number analyzed (Participants) | 70 | 71 | 141
    (all) | 10 | 12 | 22
Smoker [Count of Participants; unit: Participants] — Population: These are the baseline characteristics for the subjects who completed the study (and for whom there is outcomes data). Of the 151 subjects randomized, 4 withdrew prior to starting study med, 5 had surgery cancelled, and 1 had an intraop complication precluding any collection of outcomes data, yielding a total of 141 subjects.
  Participants
    number analyzed (Participants) | 70 | 71 | 141
    (all) | 5 | 4 | 9
COPD [Count of Participants; unit: Participants] — Chronic Obstructive Pulmonary Disease (COPD) Population: These are the baseline characteristics for the subjects who completed the study (and for whom there is outcomes data). Of the 151 subjects randomized, 4 withdrew prior to starting study med, 5 had surgery cancelled, and 1 had an intraop complication precluding any collection of outcomes data, yielding a total of 141 subjects.
  Participants
    number analyzed (Participants) | 70 | 71 | 141
    (all) | 3 | 5 | 8
Hypertension [Count of Participants; unit: Participants] — Population: These are the baseline characteristics for the subjects who completed the study (and for whom there is outcomes data). Of the 151 subjects randomized, 4 withdrew prior to starting study med, 5 had surgery cancelled, and 1 had an intraop complication precluding any collection of outcomes data, yielding a total of 141 subjects.
  Participants
    number analyzed (Participants) | 70 | 71 | 141
    (all) | 28 | 30 | 58
CHF [Count of Participants; unit: Participants] — Congestive heart failure (CHF) Population: These are the baseline characteristics for the subjects who completed the study (and for whom there is outcomes data). Of the 151 subjects randomized, 4 withdrew prior to starting study med, 5 had surgery cancelled, and 1 had an intraop complication precluding any collection of outcomes data, yielding a total of 141 subjects.
  Participants
    number analyzed (Participants) | 70 | 71 | 141
    (all) | 0 | 1 | 1
Prior MI [Count of Participants; unit: Participants] — Myocardial infarction (MI) Population: These are the baseline characteristics for the subjects who completed the study (and for whom there is outcomes data). Of the 151 subjects randomized, 4 withdrew prior to starting study med, 5 had surgery cancelled, and 1 had an intraop complication precluding any collection of outcomes data, yielding a total of 141 subjects.
  Participants
    number analyzed (Participants) | 70 | 71 | 141
    (all) | 3 | 3 | 6
BPH [Count of Participants; unit: Participants] — Benign prostatic hyperplasia (BPH) Population: These are the baseline characteristics for the subjects who completed the study (and for whom there is outcomes data). Of the 151 subjects randomized, 4 withdrew prior to starting study med, 5 had surgery cancelled, and 1 had an intraop complication precluding any collection of outcomes data, yielding a total of 141 subjects.
  Participants
    number analyzed (Participants) | 70 | 71 | 141
    (all) | 3 | 1 | 4
Prior CVA [Count of Participants; unit: Participants] — Cerebrovascular accident (CVA) Population: These are the baseline characteristics for the subjects who completed the study (and for whom there is outcomes data). Of the 151 subjects randomized, 4 withdrew prior to starting study med, 5 had surgery cancelled, and 1 had an intraop complication precluding any collection of outcomes data, yielding a total of 141 subjects.
  Participants
    number analyzed (Participants) | 70 | 71 | 141
    (all) | 3 | 2 | 5
Diabetes [Count of Participants; unit: Participants] — Population: These are the baseline characteristics for the subjects who completed the study (and for whom there is outcomes data). Of the 151 subjects randomized, 4 withdrew prior to starting study med, 5 had surgery cancelled, and 1 had an intraop complication precluding any collection of outcomes data, yielding a total of 141 subjects.
  Participants
    number analyzed (Participants) | 70 | 71 | 141
    (all) | 10 | 7 | 17
IBD [Count of Participants; unit: Participants] — Inflammatory bowel disease (IBD) Population: These are the baseline characteristics for the subjects who completed the study (and for whom there is outcomes data). Of the 151 subjects randomized, 4 withdrew prior to starting study med, 5 had surgery cancelled, and 1 had an intraop complication precluding any collection of outcomes data, yielding a total of 141 subjects.
  Participants
    number analyzed (Participants) | 70 | 71 | 141
    (all) | 20 | 16 | 36

OUTCOME MEASURES:

1. Primary Outcome: Need for Any Intermittent Catheterization Postoperatively as a Binary Outcome
Description: need for any intermittent catheterization after leaving the operating room or after initial indwelling urinary catheter (IUC) removal; subjects will be straight catheterized if the subject either 1) reports bladder discomfort, or 2) has a bladder scan for >500milliliters; or 3) has a post-void residual volume >500milliliters
Time Frame: within 0-7 days after surgery
Population: This is an intent-to-treat analysis, including all subjects who were randomized and did not withdraw prior to the intended start date of their study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Tamsulosin: Tamsulosin: Tamsulosin 0.4mg capsule orally once daily, dosed 30 minutes after dinner or before bed, starting 7 days before surgery and continuing for 0-5 days postoperatively.
- Placebo: Placebo: Placebo capsule orally once daily, dosed 30 minutes after dinner or before bed, starting 7 days before surgery and continuing for 0-5 days postoperatively.
Arm/Group | Tamsulosin | Placebo
Number analyzed (Participants) | 70 | 71
Participants | 18 | 22

2. Secondary Outcome: Need for Replacement of Indwelling Urinary Catheter as a Binary Outcome
Description: Need for replacement of an IUC after surgery or after initial removal of an IUC that was placed at the time of surgery; replacement of IUC is dictated by the institutional bladder management protocol after requiring the use of straight catheterization for 24 hours
Time Frame: within 0-7 days after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Tamsulosin | Placebo
Number analyzed (Participants) | 70 | 71
Participants | 5 | 5

3. Secondary Outcome: Time Until First Spontaneous Void
Description: time from IUC removal, last intermittent catheterization (if performed in the operating room or post-anesthesia care unit), or departure from the operating room (if no IUC placed intraoperatively) until first spontaneous void
Time Frame: within 0-7 days after surgery
Population: Time to first spontaneous void was not collected as this is not relevant clinically to diagnosis of urinary retention, and our bladder management protocol prevents unbiased collection of this data point.
Arm/Group | Tamsulosin | Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Total Number of Intermittent Catheterizations Required Per Subject
Description: total number of intermittent catheterizations required, as dictated by the institutional bladder management protocol
Time Frame: within 0-7 days after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Tamsulosin | Placebo
Number analyzed (Participants) | 70 | 71
Participants
  At least 1 catheterization | 18 | 22
  At least 2 catheterizations | 8 | 10
  greater than 2 catheterizations | 0 | 5

5. Secondary Outcome: First Post-void Residual Urine Volume
Description: The post-void residual (PVR) urine volume as measured by bedside hand-held bladder scanning immediately following the first spontaneous void
Time Frame: within 0-7 days after surgery
Population: Only includes subjects who were NOT straight-catheterized AND there were 20 additional subjects for which PVR was not recorded
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Tamsulosin | Placebo
Number analyzed (Participants) | 45 | 36
mL | 218 (167) | 154 (138)

6. Secondary Outcome: Discharge From Hospital With Indwelling Urinary Catheter
Description: Does the subject have a urinary catheter in place at the time of discharge from the hospital? This is a binary outcome measure of whether or not the subject is discharged from the hospital with an indwelling urinary catheter in place due to inadequate voiding function.
Time Frame: up to 30 days after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Tamsulosin | Placebo
Number analyzed (Participants) | 70 | 71
Participants | 0 | 0

7. Secondary Outcome: Urinary Tract Infection (UTI)
Description: Either a culture-positive UTI prior to discharge from the hospital or subject self-reported clinician-diagnosed UTI occurring within 30 days of surgery
Time Frame: up to 30 days after surgery
Population: This participant did not have urinary retention; self-reported UTI, catheter was removed on post operative day #2
Measure: Count of Participants; unit: Participants
Arm/Group | Tamsulosin | Placebo
Number analyzed (Participants) | 70 | 71
Participants | 0 | 1

8. Secondary Outcome: Hospital Length of Stay in Days
Description: Collected after the participant is discharged from the hospital, total number of consecutive days (including day of surgery) until the participant is discharged from the hospital
Time Frame: up to 30 days after surgery
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Tamsulosin | Placebo
Number analyzed (Participants) | 70 | 71
days | 6.4 (3.9) | 6.0 (3.3)

9. Secondary Outcome: Number of Participants Who Experienced Adverse Events
Description: Adverse events, systematically collected. Summary results reported here, please refer to Adverse Events section of the results record for detailed reporting.
Time Frame: treatment day 1 (7 days before surgery) until 30 days after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Tamsulosin | Placebo
Number analyzed (Participants) | 76 | 75
Participants
  Serious Adverse Events | 3 | 5
  Other Adverse Events | 10 | 8

ADVERSE EVENTS:
Time Frame: treatment day 1 (7 days before surgery) until 30 days after surgery
Description: Adverse Events were systematically collected at 3 time points (on the day of surgery from interview of the subject; during hospitalization by chart review; and 30 days after surgery from interview of the subject).
Arm/Group | Tamsulosin | Placebo
All-Cause Mortality (participants affected / at risk) | 1/76 | 0/75
Serious Adverse Events (participants affected / at risk) | 3/76 | 5/75
Other Adverse Events (participants affected / at risk) | 10/76 | 8/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tamsulosin (N=76) | Placebo (N=75)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — supratherapeutic on Lovenox leading to spontaneous rectus sheath hematoma
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 0 (0) | 1 (1) — Bleeding requiring return to the operating room
Intra-abdominal hemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Death NOS (General disorders) | 1 (1) | 0 (0) — Subject had gastric cancer, died from advanced cancer
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 (2) | 0 (0) — Ileus/SBO
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tamsulosin (N=76) | Placebo (N=75)
Blurred vision (Eye disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 6 (6) | 4 (4)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 2 (2) | 3 (3)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nervous system disorders - Other, specify (Nervous system disorders) | 1 (1) | 0 (0) — Tingling sensation
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 (1) | 1 (1) — Frequent urge to urinate
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rhinitis infective (Infections and infestations) | 0 (0) | 1 (1) — Runny nose

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-08): https://cdn.clinicaltrials.gov/large-docs/53/NCT02486653/Prot_SAP_000.pdf